CLINICAL TRIAL: NCT02987959
Title: Phase II Study of TAK-228 (MLN0128) in Soft Tissue Sarcomas With Dysregulation of the mTOR Pathway
Brief Title: Study of TAK-228 (MLN0128) in Soft Tissue Sarcomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed to accrual due to Funding Sponsor withdrawing support due to low accrual
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAR-081
Record Dates: First submitted 2016-12-02; First posted 2016-12-09 (Estimated); Results first posted 2021-02-24 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-09

CONDITIONS: Soft-tissue Sarcoma
Keywords: TAK-228; MLN0128; mTOR
MeSH Terms: conditions — Sarcoma | interventions — sapanisertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAK-228 treatment (Experimental): Patients with complex genomic sarcomas exhibiting PI3K pathway dysregulation will be treated with TAK-228
  Interventions: Drug: TAK-228

INTERVENTIONS:
Drug: TAK-228 — TAK-228 is a novel, highly selective, orally bioavailable adenosine 5' triphosphate (ATP)-competitive inhibitor of the serine/threonine kinase referred to as the mechanistic target of rapamycin (mTOR). TAK-228 (formerly INK128) targets 2 distinct mTOR complexes, mTOR complex 1 (mTORC1) and mTOR complex 2 (mTORC2).
  Other Names: MLN0128

SUMMARY:
This is an open-label phase II study of TAK-228 for patients ≥ 18 years of age with complex genomic sarcomas exhibiting Phosphoinositide-3 Kinase (PI3K) pathway dysregulation. Patients must have surgically unresectable or metastatic disease that is refractory to at least one prior line of therapy (not including neoadjuvant or adjuvant therapy in a curative setting). Patients disease must also have evidence of progression prior to enrollment. The purpose of this study is to determine the antitumor activity in this group of patients. Patients must meet all eligibility criteria as detailed in section 10. A total of up to 33 patients will be included in the study. Patients will undergo screening evaluations to determine eligibility within 28 days of the first dose. All patients will be required to submit baseline tumor samples for analysis. Patients who have had their tumors tested commercially for PI3K/ AKT/mechanistic Target of Rapamycin (mTOR) alterations will be assessed on a case by case basis for eligibility and for determination as to whether additional tissue is required.

TAK-228 will be administered orally at 3 mg daily for a 21 day cycle. Clinical and laboratory assessments will be made on day 1 of each cycle. Disease will be assessed by comparing unidimensional tumor measurements on pre and peritreatment imaging (CT or MRI) after weeks 6, 12, 18 and every 12 weeks thereafter. Response will be assessed according to RECIST 1.1. Therapy will continue until disease progression or unacceptable toxicity or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* This trial has two step inclusion criteria.

Step 1 Inclusion Criteria

1. Male or female patients 18 years or older.
2. Patients must have a diagnosis of a locally advanced or metastatic sarcoma that is progressing. The following subtypes (considered genomically complex) will be eligible: leiomyosarcoma (well differentiated or poorly differentiated), undifferentiated pleomorphic sarcoma, myxofibrosarcoma, pleomorphic rhabdomyosarcoma, pleomorphic liposarcoma, malignant peripheral nerve sheath tumor, angiosarcoma or extraskeletal osteosarcoma. Other potentially genomically complex Soft Tissue Sarcomas (STS) subtypes may be included on a case-by-case basis after discussion with the principal investigator.
3. Measurable disease by RECIST 1.1 criteria (at least one target lesion outside of previous radiation fields or progressed within a previous radiation field), described in detail in section 15.
4. Progression of disease by radiographic imaging (10% increase in size by RECIST v1.1 within 6 months of registration) or presence of new lesions.
5. Must have received at least 1 prior systemic therapy for advanced disease (does not include adjuvant/neoadjuvant therapy in a curative setting).
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
7. Adequate contraception as follows:

   For women:

   Postmenopausal for at least 1 year before the screening visit, OR Surgically sterile, OR If they are of childbearing potential, agree to practice 1 effective method of contraception, and 1 additional (barrier) method, at the same time, from the time of signing the informed consent through 90 days (or longer, as mandated by local labeling [eg. United Surgical Partners Internationals (USPI), Summary of Product Characteristics (SmPC), etc;]) after the last dose of study drug OR agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient (Periodic abstinence [e.g, calendar, ovulation, symptothermal, postovulation methods] and withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)

   Highly effective methods:

   Intra-uterine devices (IUD) Hormonal (birth control pills/oral contraceptives, injectable contraceptives, contraceptive patches, or contraceptive implants)

   Other effective Methods:

   Latex Condoms Diaphragm with spermicide; Cervical cap;Sponge

   For men, even if surgically sterilized (ie, status post-vasectomy), they must:

   Agree to practice highly effective barrier contraception during the entire study treatment period and through 120 days after the last dose of study drug, OR agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient (Periodic abstinence [e.g, calendar, ovulation, symptothermal, postovulation methods for the female partner] and withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)

   Agree not to donate sperm during the course of this study or 120 days after receiving their last dose of study drug
8. Screening clinical laboratory values as specified below:

   a) Bone marrow reserve consistent with: i. absolute neutrophil count (ANC) ≥ 1.5 x 10(9)/L; ii. platelet count ≥ 100 x 10(9)/L; iii. hemoglobin ≥ 9 g/dL without transfusion within 1 week preceding study drug administration b) Hepatic: i. total bilirubin ≤ 1.5 x upper limit of normal (ULN), ii. transaminases (Aspartate aminotransferase/Serum Glutamic Oxaloacetic Transaminase (AST/SGOT) and Alanine aminotransferase/Serum Glutamic Pyruvic Transaminase (ALT/SGPT) ≤ 2.5 x ULN (≤ 5 x ULN if liver metastases are present); c) Renal: creatinine clearance ≥ 50 mL/min based either on Cockcroft-Gault estimate or based on urine collection (12 or 24 hour); d) Metabolic: i. Glycosylated hemoglobin (HbA1c) ≤ 7.0%, ii. fasting serum glucose ≤ 130 mg/dL iii. fasting triglycerides ≤ 300 mg/dL
9. Ability to swallow oral medications.
10. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
11. Patients who have a history of brain metastasis are eligible for the study provided that all the following criteria are met:

    1. Brain metastases which have been treated
    2. No evidence of disease progression for ≥ 3 months or hemorrhage after treatment
    3. Off-treatment with dexamethasone for 4 weeks before administration of the first dose of TAK-228
    4. No ongoing requirement for dexamethasone or anti-epileptic drugs

Step 2 Inclusion Criteria: Must be met after meeting step1inclusion and exclusion criteria.

1. Tumor must have dysregulation of the PI3K/AKT/mTOR pathway. For the purposes of this study, patients must have either PTEN protein or genomic loss, or phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha (PIK3CA)/ Phosphatase and tensin homolog (PTEN) mutation. Patients must be willing to provide sufficient archival tissue. If this is not available fresh tumor for biopsy is required. In the event that a patient has had tumor analyzed for PTEN/PIK3CA status through commercial means, their eligibility and need for additional tissue will be determined on a case by case basis by the principle investigator.

Exclusion Criteria:

* Step 1 Exclusion Criteria

  1. Any clinically significant co-morbidities, such as uncontrolled pulmonary disease, active central nervous system disease, active infection, or any other condition that could compromise the patient's participation in the study.
  2. Known human immunodeficiency virus infection.
  3. Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection.
  4. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
  5. Diagnosed or treated for another malignancy within 2 years before administration of the first dose of study drug, or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
  6. Breast feeding or pregnant.
  7. Manifestations of malabsorption due to prior gastrointestinal (GI) surgery, GI disease, or for an unknown reason that may alter the absorption of TAK-228. In addition, patients with enteric stomata are also excluded.
  8. Treatment with any investigational products, radiation therapy, surgery, tumor embolization, chemotherapy or immunotherapy within 21 days before the first dose of the study drug. For biologic or hormonal therapy treatment within 14 days or five half-lives of a drug (whichever is longer) before the first dose of study drug.
  9. History of any of the following within the last 6 months before administration of the first dose of the drug:

     1. Ischemic myocardial event, including angina requiring therapy and artery revascularization procedures
     2. Ischemic cerebrovascular event, including transient ischemic attack and artery revascularization procedures
     3. Requirement for inotropic support (excluding digoxin) or serious (uncontrolled) cardiac arrhythmia (including atrial flutter/fibrillation, ventricular fibrillation or ventricular tachycardia)
     4. Placement of a pacemaker for control of rhythm
     5. New York Heart Association (NYHA) Class III or IV heart failure
     6. Pulmonary embolism
  10. Significant active cardiovascular or pulmonary disease including:

      1. Uncontrolled hypertension (i.e., systolic blood pressure >180 mm Hg, diastolic blood pressure >95 mm Hg). Use of anti-hypertensive agents to control hypertension before Cycle1 Day 1 is allowed.
      2. Pulmonary hypertension
      3. Uncontrolled asthma or O2 saturation < 90% by arterial blood gas analysis or pulse oximetry on room air
      4. Significant valvular disease; severe regurgitation or stenosis by imaging independent of symptom control with medical intervention, or history of valve replacement
      5. Medically significant (symptomatic) bradycardia
      6. History of arrhythmia requiring an implantable cardiac defibrillator
      7. Baseline prolongation of the rate-corrected QT interval (QTc) (e.g., repeated demonstration of QTc interval >480 milliseconds, or history of congenital long QT syndrome, or torsades de pointes)
  11. Poorly controlled diabetes mellitus defined as glycosylated hemoglobin (HbA1c) >7% ; patients with a history of transient glucose intolerance due to corticosteroid administration or gestational diabetes may be enrolled in this study if all other inclusion/exclusion criteria are met.
  12. Treatment with strong inhibitors and/or inducers of cytochrome P450 (CYP) 3A4, CYP2C19 or CYP2C9 within 1 week preceding the first dose of study drug.
  13. Patients receiving systemic corticosteroids (either IV or oral steroids, excluding inhalers or low-dose hormone replacement therapy) within 1 week before administration of the first dose of study drug.
  14. Daily or chronic use of a proton pump inhibitor (PPI) and/or having taken a PPI within 7 days before receiving the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2020-07-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAK-228 Treatment
Started | 6
Completed | 0
Not Completed | 6
Not completed — Grantor stopped supply of drugs | 6

BASELINE CHARACTERISTICS:
Arm/Group | TAK-228 Treatment
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 53 [27 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
Tumor type [Count of Participants; unit: Participants]
  Leiomyosarcoma | 4
  Extraskeletal osteosarcoma | 1
  Soft tissue sarcoma | 1

OUTCOME MEASURES:

1. Primary Outcome: The Progression Free Survival Rate With TAK-228 in Sarcoma Patients With PI3K/AKT/mTOR Pathway Dysregulation
Description: Progression free rate will be determined by determining the number of patients with complete response, partial response and stable disease
Time Frame: 12 weeks post-treatment
Population: Insufficient number of patients accrued for a meaningful analysis. No data collected from any participant.
Arm/Group | TAK-228 Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: The Rate of Toxicity of TAK-228 in This Patient Population as Per Common Terminology Criteria for Adverse Events (CTCAE)v4.03 Criteria.
Description: Toxicity will be assessed by calculating number of participants experiencing adverse events as per CTCAEv4.03 criteria
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-228 Treatment
Number analyzed (Participants) | 6
Participants | 6

3. Secondary Outcome: The Objective Response Rate (ORR) of TAK-228 in This Patient Population.
Description: Objective response rate will be defined as patients with complete response and partial response. As per RECIST v1.1 guidelines, complete response is defined as the disappearance of all measurable lesions, and partial response is defined as >=30% decrease in sum of diameters of target lesions compared to the baseline sum of diameters.
Time Frame: upto 4 years
Population: Insufficient number of patients accrued for a meaningful analysis. No data collected from any participant.
Arm/Group | TAK-228 Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression Free Survival in This Patient Population.
Description: Progression Free Survival, defined as the time from initiation of treatment until disease progression will be calculated.
Time Frame: upto 4 years
Population: Insufficient number of patients accrued for a meaningful analysis. No data collected from any participant.
Arm/Group | TAK-228 Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival Rate in This Patient Population
Description: Overall Survival, defined as the time from initiation of treatment until death from any cause will be calculated.
Time Frame: upto 4 years
Population: Insufficient number of patients accrued for a meaningful analysis. No data collected from any participant.
Arm/Group | TAK-228 Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | TAK-228 Treatment
All-Cause Mortality (participants affected / at risk) | 4/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAK-228 Treatment (N=6)
Acute kidney injury (Renal and urinary disorders) | 1 (1) — Grade 3 acute kidney injury
Intractable nausea and vomiting (Gastrointestinal disorders) | 1 (1) — Patient was hospitalized after 4 days of nausea and vomiting with some loose stools
Septic arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 3 septic arthritis in the knee
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAK-228 Treatment (N=6)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Taste alteration (Gastrointestinal disorders) | 1 (1) — Gastrointestinal disorders - Other
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Pain (General disorders) | 2 (2)
Edema (General disorders) | 1 (1) — Edema limbs
Fever (General disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) — Myalgia
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Back pain
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) — Generalized muscle weakness
Right hip cramps (Musculoskeletal and connective tissue disorders) | 1 (1) — Musculoskeletal and connective tissue disorder - Other, specify
Dizziness (Nervous system disorders) | 2 (2) — Dizziness
Headache (Nervous system disorders) | 1 (1) — Headache
Syncope (Nervous system disorders) | 1 (1) — Syncope
Tremor (Nervous system disorders) | 1 (1) — Tremor
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Dyspnea
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Cough
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Epistaxis
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Nasal congestion
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Shortness of breath
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) — Rash maculo-papular
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (2) — Itching and hives
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) — Dry skin
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) — Pruritus
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) — Light headedness
Palpitations (Cardiac disorders) | 1 (1) — Palpitations
Infections and infestations - Other, specify (Infections and infestations) | 2 (2) — Infection
Investigations - Other, specify (Investigations) | 2 (2) — Discomfort anterior portion right leg Sweats
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) — Activated partial thromboplastin time prolonged
Alanine aminotransferase increased (Investigations) | 1 (1) — Alanine aminotransferase increased
Weight loss (Investigations) | 1 (1) — Weight loss
White blood cell decreased (Investigations) | 1 (1) — White blood cell decreased
Anorexia (Metabolism and nutrition disorders) | 1 (1) — Anorexia
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) — Hyperglycemia
Proteinuria (Renal and urinary disorders) | 1 (1) — Proteinuria
Anemia (Blood and lymphatic system disorders) | 1 (1) — Anemia
Eye disorders - Other, specify (Eye disorders) | 1 (1) — Eye itching
Wound complication (Injury, poisoning and procedural complications) | 1 (1) — Wound right knee
Depression (Psychiatric disorders) | 1 (1) — Depression

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT02987959/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT02987959/ICF_001.pdf